CLINICAL TRIAL: NCT06187818
Title: Study of Crocin on Cardiac Function Protection in Patients With Breast Cancer Undergoing Neoadjuvant Chemotherapy Based on Color Doppler Ultrasound Combined With Myocardial Zymogram
Brief Title: Follow up Study of Crocin on Cardiac Function Protection in Patients With Breast Cancer Undergoing Neoadjuvant Chemotherapy Based on Color Doppler Ultrasound Combined With Myocardial Zymogram
Status: Active, not recruiting | Type: Observational
Sponsor: Mei Zhang (Other)
Responsible Party: Sponsor-Investigator, Mei Zhang, Deputy chief physician, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: 2023006
Record Dates: First submitted 2023-12-17; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — crocin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- experience group 1: Take 4 total glucosides of crocin tablets (Ruiyang Pharmaceutical Co., Ltd.) 3 times a day for 8 days (the day before chemotherapy) during each chemotherapy.Previous history of heart disease.
  Interventions: Drug: Crocin
- experience group 2: Take 4 total glucosides of crocin tablets (Ruiyang Pharmaceutical Co., Ltd.) 3 times a day for 8 days (the day before chemotherapy) during each chemotherapy.No previous heart disease.
  Interventions: Drug: Crocin
- Control group 1: Did not take crocine tablets during chemotherapy.Previous history of heart disease.
- Control group 2: Did not take crocine tablets during chemotherapy.No previous heart disease.

INTERVENTIONS:
Drug: Crocin — According to the patient's condition, tolerance level, and personal preference, the dosage of medication was selected. During chemotherapy, the total anthocyanin tablets were divided into an experimental group (experimental group 1 and experimental group 2 based on previous heart disease) and a control group (control group 1 and control group 2 based on previous heart disease), 30 cases in each group [experimental group: taking saffron total glycoside tablets for 8 days during each chemotherapy period (starting from the day before chemotherapy), 4 tablets/time, 3 times a day; control group: not taking saffron total glycoside tablets during chemotherapy period]
  Groups: experience group 1; experience group 2

SUMMARY:
Foreign data show that: 1807 tumor patients were followed up for 7 years, 33% of them died of heart disease and 51% of them died of the tumor itself. In China, the number of cancer patients undergoing chemotherapy is increasing rapidly every year. How to protect the heart of chemotherapy patients from the damage of chemotherapy drugs (especially anthracyclines) is a problem that clinicians must face.In order to further confirm the clinical efficacy and value of saffron total glycosides tablets in the protection of central function of breast cancer neoadjuvant patients with anthracycline based chemotherapy scheme, the project plans to follow up and observe the research of saffron total glycosides on the protection of cardiac function of breast cancer neoadjuvant patients with chemotherapy based on cardiac color ultrasound combined with myocardial zymography, and randomly group to confirm the effectiveness of saffron total glycosides tablets on cardiac protection, Based on the clinical observation and research on the effect of traditional Chinese medicine on the cardiotoxicity of anthracycline drugs, confirm its efficacy, explore the mechanism of cardiac protection, and explore the drug use method of synergism and toxicity reduction of anthracycline drugs in combination with this active ingredient.

DETAILED DESCRIPTION:
At present, the commonly used anthracycline antineoplastic drugs in clinic include daunorubicin, doxorubicin, epirubicin, pirarubicin, idabicin, pentarubicin and mitoxantrone, among which doxorubicin is one of the most commonly used antineoplastic drugs. However, anthracyclines have dose dependent and cumulative cardiotoxicity. In patients receiving doxorubicin (DOX) treatment, nearly 10% of patients will have cardiac complications after stopping chemotherapy for nearly 10 years, and its cardiac toxicity may even threaten life, which limits its clinical application.

Crocus sativus glycoside, as the main active ingredient of Crocus sativus L., has a wide range of pharmacological effects, and it has a good effect on cardiovascular system.

Based on the clinical observation and research on the effect of traditional Chinese medicine on the cardiotoxicity of anthracycline drugs, confirm its efficacy, explore the mechanism of cardiac protection, and explore the drug use method of synergism and toxicity reduction of anthracycline drugs in combination with this active ingredient. In this study, 120 patients with breast cancer undergoing neoadjuvant chemotherapy (including anthracycline) were randomly enrolled, and the cardiac baseline assessment was done. The clinical efficacy of crocin in protecting heart function of breast cancer patients undergoing neoadjuvant chemotherapy was evaluated according to clinical symptoms, cardiac color ultrasound, electrocardiogram and myocardial enzyme spectrum, To further verify the clinical application value and social and economic benefits of saffron, the heart protecting active ingredient in saffron, in the aspect of heart protection in neoadjuvant chemotherapy for breast cancer, and further promote the use and broaden the clinical application range of traditional Chinese medicine. Prevention is more important than treatment, which is in line with the national concept of "preventing disease" of traditional Chinese medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with breast cancer aged ≥ 20 years and ≤ 80 years, with informed consent and meeting the treatment standard of neoadjuvant chemotherapy scheme.
2. Patients who plan to receive neoadjuvant chemotherapy based on anthracycline drugs (such as erythromycin, doxorubicin, epirubicin, pyranomycin, idabicin, pentorubicin, and mitoxantrone).
3. No treatment for breast cancer before enrollment, such as chemotherapy, targeted therapy and endocrine therapy.
4. All patients underwent coarse needle biopsy of breast tumors (axillary lymph node biopsy is required for suspected axillary lymph node metastasis) to determine the status of ER, PR, HER-2, and Ki-67.
5. All patients have normal lung function, liver and kidney function.

Exclusion Criteria:

1. Cases that do not cooperate and are unwilling to sign informed consent forms.
2. Antitumor therapy, hormone replacement therapy and other breast cancer related treatments were performed before enrollment.
3. Merge any other malignant tumors.
4. Patients with poor image quality in echocardiography.
5. Continuous atrial fibrillation and severe arrhythmia affect ultrasound data collection and analysis.
6. Patients with active infections, a history of HIV, or chronic hepatitis B or C.
7. Patients with abnormal lung function or liver and kidney function.
8. Patients with hemorrhagic diseases.
9. Patients taking other heart protection traditional Chinese patent medicines and simple preparations.
10. Participated in other clinical researchers in the past 3 months.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients with neoadjuvant chemotherapy based on anthracycline drugs who were hospitalized in the breast surgery department of Shandong Qianfoshan Hospital from the time when the ethical approval document was obtained to December 2024.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac ultrasound LVEF, GLS | December 2024
  LVEF and GLS levels measured by echocardiography before and after treatment (within and between groups).

SECONDARY OUTCOMES:
Abnormal rate of electrocardiogram | December 2024
  Comparison of abnormal electrocardiogram rates before and after treatment (within and between groups).
Overall radial strain of the heart | December 2024
  Overall radial strain measured by ultrasound before and after treatment (intra group and inter group).
Cardiac asynchrony index | December 2024
  Cardiac asynchrony index before and after treatment (within and between groups).
myocardial enzymes | December 2024
  Comparison of myocardial enzyme spectrum results before and after treatment (within and between groups).
Symptoms of cardiac discomfort | December 2024
  The frequency and duration of chest tightness, chest pain, and palpitations.

CONTACTS AND LOCATIONS:
Overall Officials: Guoming Liu, master, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University (Qianfo Mountain Hospital); Zhanpeng Zhao, master, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University (Qianfo Mountain Hospital); Xinlei Zhang, master, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University (Qianfo Mountain Hospital); Yonghao Li, master, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University (Qianfo Mountain Hospital); Xuena Zhao, master, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University (Qianfo Mountain Hospital)
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital in Shandong Province), Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided